CLINICAL TRIAL: NCT07356934
Title: The Effect of a Health Belief Model-Based Web Education Program on Self-Efficacy and Home Accident Awareness Among Mothers of Children Aged 0-3 in Family Health Centers: A Randomized Controlled Experimental Study
Brief Title: Health Belief Model-Based Web Education for Preventing Home Accidents in Mothers of Children Aged 0-3
Acronym: HBM-HAWE
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ataturk University (Other)
Responsible Party: Principal Investigator, Şeyda Uzunlu, PhD Candidate, Department of Public Health Nursing, Ataturk University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: B.30.2.ATA.0.01.00/394; TDK-2025-16163 (Other Grant/Funding Number: Atatürk University)
Record Dates: First submitted 2026-01-13; First posted 2026-01-21 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Accident Prevention; Wounds and Injuries; Accidental Falls
Keywords: Health Belief Model; Web-Based Education; Mothers; Self-Efficacy; Awareness
MeSH Terms: conditions — Wounds and Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HBM-Based Web Education Program (Experimental): Participants receive usual care plus a Health Belief Model (HBM)-based web education program on prevention of home accidents in children aged 0-3 years. The program is delivered via a dedicated website over 3 months and includes six structured modules (perceived susceptibility, perceived severity, perceived benefits, perceived barriers, and self-efficacy). The intervention is supported by WhatsApp reminder messages, an interactive "Ask Us" feature, and two Zoom meetings during follow-up.
  Interventions: Behavioral: HBM-Based Web Education for Home Accident Prevention
- Usual Care (Control) (No Intervention): Participants receive usual care provided by the Family Health Center. They do not receive the HBM-based web education program during the study period. After completion of post-test data collection, participants in this group will be provided with the educational booklet containing the same information as the website.

INTERVENTIONS:
Behavioral: HBM-Based Web Education for Home Accident Prevention — A structured Health Belief Model (HBM)-based web education program designed to improve mothers' self-efficacy and awareness regarding prevention of home accidents in children aged 0-3 years. The intervention is delivered via a dedicated website over 3 months and consists of six modules covering perceived susceptibility, severity, benefits, barriers, and self-efficacy. Educational content includes visual materials and videos. The program is supported by WhatsApp reminder messages, an interactive "Ask Us" feature for participant questions, and two Zoom meetings during follow-up.
  Arms: HBM-Based Web Education Program

SUMMARY:
This randomized controlled experimental study evaluates the effect of a Health Belief Model (HBM)-based web education program on preventing home accidents among mothers of children aged 0-3 years registered in a Family Health Center in Erzurum, Türkiye. Unintentional injuries such as falls, burns, poisoning, choking/aspiration, and cutting/piercing injuries are common in early childhood and often occur in the home environment. Mothers play a critical role in recognizing home hazards and implementing preventive safety behaviors.

Participants will be randomly assigned to either an intervention group (HBM-based web education) or a control group (usual care). The intervention includes a structured web-based education program delivered over three months, supported by reminder messages via WhatsApp, interactive communication through an "Ask Us" option, and two Zoom meetings during the follow-up period. Outcomes will be measured using the General Self-Efficacy Scale and the Mother Home Accidents Awareness Scale. Baseline data will be collected through face-to-face interviews before the intervention, and post-test data will be collected at the 6th month. The study aims to determine whether HBM-based digital education improves maternal self-efficacy and awareness regarding home accident prevention.

DETAILED DESCRIPTION:
This study evaluates a theory-driven digital education intervention designed to improve maternal preventive behaviors related to early childhood home safety. The intervention is grounded in the Health Belief Model (HBM), which explains preventive health actions through perceived susceptibility, perceived severity, perceived benefits, perceived barriers, and self-efficacy. In the context of home accidents, the model is used to strengthen risk perception, increase motivation for adopting safety practices, reduce perceived obstacles to prevention, and enhance caregiver confidence in implementing protective behaviors.

The intervention is delivered through a structured web-based education platform tailored for mothers of young children. The content is organized into sequential modules mapped directly to HBM constructs. Educational materials are designed to support learning through multimodal delivery (written content, visuals, and videos) and to encourage practical application of safety behaviors in the home environment. In addition to asynchronous web learning, the intervention incorporates reinforcement and engagement strategies, including periodic reminder messaging and interactive communication options that allow participants to ask questions and receive feedback. Scheduled online meetings are included to support understanding, troubleshoot barriers, and promote sustained participation.

Participants are assigned to study groups using a random allocation approach. The trial uses a pre-test/post-test structure to quantify changes over time and to compare outcomes between study arms. Data analysis will follow a structured statistical plan, including descriptive summarization and group comparisons, with reliability checks for the measurement tools used in the study. Ethical approvals and institutional permissions have been obtained, and all study procedures are conducted in accordance with applicable ethical standards for research involving human participants.

ELIGIBILITY:
Inclusion Criteria:

Female participants who are mothers of at least one child aged 0-3 years

Registered at the participating Family Health Center

Aged 18-49 years

Able to read and write sufficiently to understand study materials and complete questionnaires

Able to communicate effectively and follow study instructions

Has no physical, cognitive, or mental condition that would prevent participation in the education program or completion of assessments

Has access to the internet via a smartphone, tablet, or computer

Willing to participate in the study and able to provide written informed consent

Exclusion Criteria:

Relocation to another city or region during the study period

Development of any medical, psychological, or social condition that prevents continued participation

Inability to complete follow-up assessments for any reason

Withdrawal of consent or voluntary withdrawal from the study at any time

Ages: 18 Years to 49 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 140 (Estimated)
Dates: Start 2025-11-02 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Mother Home Accidents Awareness Score | Baseline (pre-test) and 6 months (post-test)
  Home accident awareness will be assessed using the Mother Home Accidents Awareness Scale, a 55-item instrument rated on a 5-point Likert scale. The scale includes four domains: fall awareness, burn awareness, poisoning awareness, and choking/drowning awareness, as well as cutting/piercing injury awareness. Total scores range from 55 to 275, with higher scores indicating greater home accident awareness (better outcome).
General Self-Efficacy Score | Baseline (pre-test) and 6 months (post-test)
  General self-efficacy will be assessed using the General Self-Efficacy Scale. Total scores range from 17 to 85, with higher scores indicating greater self-efficacy (better outcome). Items designated by the scale are reverse-scored according to standard scoring procedures.

CONTACTS AND LOCATIONS:
Locations (1):
- Maksut Efendi Family Health Center (ASM), Erzurum, Yakutiye, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Janz NK, Becker MH. The Health Belief Model: a decade later. Health Educ Q. 1984 Spring;11(1):1-47. doi: 10.1177/109019818401100101. PMID 6392204
- [Background] Cummings KM, Jette AM, Rosenstock IM. Construct validation of the health belief model. Health Educ Monogr. 1978 Winter;6(4):394-405. doi: 10.1177/109019817800600406. PMID 299611
- [Background] Bandura A. Self-efficacy: toward a unifying theory of behavioral change. Psychol Rev. 1977 Mar;84(2):191-215. doi: 10.1037//0033-295x.84.2.191. No abstract available. PMID 847061